CLINICAL TRIAL: NCT02673086
Title: Could the Retroclavicular Block Alternative for Ultrasound-guided Infraclavicular Block: A Prospective Randomized Controlled Trial
Brief Title: Retroclavicular Versus Coracoid Approach for Infraclavicular Brachial Plexus Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Antalya Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: AntalyaTRH 010
Record Dates: First submitted 2016-01-19; First posted 2016-02-03 (Estimated); Last update posted 2017-06-19 (Actual); Status verified 2016-08

CONDITIONS: Disorder of Upper Extremity
Keywords: retroclavicular approach; coracoid approach; ultrasound; upper limb surgery; needle visibility; infraclavicular brachial plexus block

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- coracoid approach (Active Comparator): Patients in this group will be randomized to receive an coracoid approach to Ultrasound Guided Infraclavicular Brachial Plexus Nerve Block .
  Interventions: Other: coracoid approach
- retroclavicular approach (Active Comparator): Patients in this group will be randomized to receive an retroclavicular approach to Ultrasound Guided Infraclavicular Brachial Plexus Nerve Block .
  Interventions: Other: retroclavicular approach

INTERVENTIONS:
Other: coracoid approach — Coracoid approach for ultrasound guided infraclavicular brachial plexus block
  Arms: coracoid approach
Other: retroclavicular approach — retroclavicular approach for ultrasound guided infraclavicular brachial plexus block
  Arms: retroclavicular approach

SUMMARY:
The primary aim of this study is to compare needle tip visibility between the coracoid approach and retroclavicular approach for infraclavicular brachial plexus block in patients undergoing elective upper limb surgery. Secondary aim is to investigate the differences between the two groups in the needle shaft visibility, sensorial block success rate, block performance time, block performance related pain, motor block success rate, surgical success rate, complications, patient satisfaction, use of supplemental local anesthetic, use of analgesic.

DETAILED DESCRIPTION:
Infraclavicular blocks are performed with different approaches. Infraclavicular block is usually traditionally performed at coracoid approach. Different approaches has been described for this block such as vertical approach. This study evaluated the effectiveness, safety and feasibility of a retroclavicular brachial plexus block as compared with traditionally coracoid approach for infraclavicular brachial plexus block. 100 patients scheduled for elective upper limb surgery were recruited and randomized into two groups: Coracoid approach for infraclavicular block (Group I), retroclavicular approach for infraclavicular block (Group R). Sensory block, adverse effects and complications were evaluated and recorded every 10 minutes until 30min after local anesthetic injection.Success rate of each nerve sensory block, complications, rate of satisfaction, rate of failure and incidence rate of adverse effects, the needle tip and shaft visibility, procedure time,duration of the block's effect, use of supplemental local anesthetic, use of analgesic.are compared with both groups.

ELIGIBILITY:
Inclusion Criteria:

* patients who undergo elective forearm or hand surgery under infraclavicular brachial plexus block
* American Society of Anesthesiologists class 1 to 3
* Ability to consent

Exclusion Criteria:

* History of allergic reaction to local anaesthetics
* Peripheral neuropathy
* Renal or hepatic insufficiency
* Coagulation disorders

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-12; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Needle visibility | 10 minutes after the needle inserted the skin
  To assess the needle visibility will be reviewed by two anesthesiologists using a 5-point Likert scale.

SECONDARY OUTCOMES:
Technique duration | Time required in seconds for the block completion (10 minutes)
  Number of seconds needed to complete the block, from time the first insertion of the blocking needle to its removal.
Patient satisfaction using a visual analogue scale | Assessed 48 hours after the block
  Using a visual analogue scale , patients will quantify their satisfaction with the retroclavicular coracoid technique.
Surgical success rate | 6 hours after the block
  Surgical success is defined as no requirement for additional local anesthetic and the use of intravenous analgesic, rescue blocks, or general anesthesia during the surgery.
supplemental analgesic use | 90 minutes after block completion
  the need for additional intravenous analgesic
complications such as pneumothorax, hemothorax, intraarterial injection, intravenous injection | 24 hours
  Patients are asked about possible complications and all the patients studied is evaluated by performing bedside ultrasound examinations of the chest before discharge.
motor block success rate | Assessed 40 minutes after block completion
  Motor function is evaluate for flexion of the elbow, opposition of the thumb, and adduction of the thumb based on a three point scale (0 = normal strength, 1 = paresis, 2 = paralysis)
Success Rate of the sensorial Block | Assessed 30 minutes after block completion
  Sensory assessments are performed every 5 minutes after needle removal for 30 minute in the regions of the radial, median, ulnar, musculocutaneous of the forearm based on a three point scale with cold test ( 0: normal sensation, 1:analgesia, 2: anesthesia).
Block performance related pain | 10 minutes after the needle inserted the skin
  Block performance related pain is evaluated with a verbal rating scale score after the removel of the needle.

CONTACTS AND LOCATIONS:
Overall Officials: Nılgun Kavrut Ozturk, MD, Study Director — Antalya Training and Research Hospital
Locations (1):
- Antalya Training and Research Hospital, Department of Anesthesiology and Reanimation, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kavrut Ozturk N, Kavakli AS. Comparison of the coracoid and retroclavicular approaches for ultrasound-guided infraclavicular brachial plexus block. J Anesth. 2017 Aug;31(4):572-578. doi: 10.1007/s00540-017-2359-6. Epub 2017 Apr 18. PMID 28421316